CLINICAL TRIAL: NCT03695510
Title: Afatinib and Pembrolizumab for Recurrent or Metastatic Head and Neck Squamous Cell Carcinoma, A Single-Arm, Phase II Study (ALPHA Study)
Brief Title: Afatinib and Pembrolizumab for Head and Neck Squamous Cell Carcinoma (ALPHA Study)
Acronym: ALPHA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201803071MIPD
Record Dates: First submitted 2018-10-01; First posted 2018-10-04 (Actual); Last update posted 2022-04-21 (Actual); Status verified 2022-04

CONDITIONS: Head and Neck Neoplasms
Keywords: head and neck cancer,Immunotherapy
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Afatinib; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Study arm (Experimental): afatinib + pembrolizumab
  Interventions: Drug: Afatinib Oral Tablet; Drug: Pembrolizumab Injection

INTERVENTIONS:
Drug: Afatinib Oral Tablet — 40mg oral, daily, continuously
  Other Names: Giotrif
Drug: Pembrolizumab Injection — 200mg, intra-venous injection, every 3 weeks, for 35 cycles
  Other Names: Keytruda

SUMMARY:
The primary objectives of the trial is to examine the toxicities and efficacies of afatinib and pembrolizumab for recurrent and/or metastatic head and neck squamous cell carcinoma.

DETAILED DESCRIPTION:
It is a single arm, phase II, single center, prospective, open label clinical trial.

ELIGIBILITY:
Inclusion criteria

1. Histologically confirmed squamous cell carcinoma of oral cavity, oropharynx, hypopharynx, or larynx.
2. The recurrent disease is not suitable for curative surgery or definitive chemoradiation, and/or metastatic diseases which are not amenable to surgery and/or curative radiotherapy.
3. Tumor progression or recurrence within 6 months of last dose of platinum therapy in the adjuvant (ie with radiation after surgery), primary (ie, with radiation), recurrent, or metastatic setting. Clinical progression after platinum therapy is an allowable event for entry and is defined as progression of a lesion at least 10 mm in size that is amenable to caliper measurement (eg superficial skin lesion as per RECIST 1.1) or a lesion that has been visualized and photographically recorded with measurements and shown to have progressed.
4. Measurable disease according to RECIST 1.1. Lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.
5. Age ≥ 20 years
6. ECOG performance status: ≤ 2
7. Adequate organ function
8. Recovered from any previous therapy related toxicity to ≤Grade 1 at study entry (except for stable sensory neuropathy ≤Grade 2 and alopecia)
9. Agree to take biopsy before and during the treatment
10. The participant (or legally acceptable representative if applicable) provides written informed consent for the trial.
11. Female subject of childbearing potential should have a negative urine pregnancy test within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
12. Female subjects of childbearing potential must be willing to use an adequate method of contraception, for the course of the study through 60 days after the last dose of study medication.

    Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.
13. Male subjects of childbearing potential must agree to use an adequate method of contraception, starting with the first dose of study therapy through 150 days after the last dose of study therapy.

Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.

3.3.3 Exclusion criteria

1. Nasopharyngeal carcinoma or nasal cavity malignancies other than HNSCC
2. Concurrent malignancies other than HNSCC
3. Prior exposure to anti-PD-1, anti-PD-L1, anti-CTLA-4, or other immune checkpoint inhibitors
4. Prior exposure to gefitinib, erlotinib, afatinib, osimertinib, or other known EGFR TKI inhibitors
5. Has a known history of Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive) or known active Hepatitis C virus (defined as positive anti-HCV) infection.
6. Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
7. Has an active infection requiring systemic therapy 14 days before signing informed consent.
8. Has received prior radiotherapy within 2 weeks of start of study treatment. Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (≤2 weeks of radiotherapy) to non-CNS disease.
9. Major surgery within 4 weeks before starting study treatment or scheduled for surgery during the projected course of the study.
10. History or presence of clinically relevant cardiovascular abnormalities such as uncontrolled hypertension, congestive heart failure NYHA classification of ≥ 3, unstable angina or poorly controlled arrhythmia as determined by the investigator. Myocardial infarction within 6 months prior to randomisation.
11. Has known history of pneumonitis requiring steroids, or any evidence of active, non-infectious pneumonitis, or other known interstitial lung disease
12. Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
13. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment. Topical or inhaled steroids is not considered as systemic treatment.
14. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
15. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
16. Any history of or concomitant condition that, in the opinion of the Investigator, would compromise the patient's ability to comply with the study or interfere with the evaluation of the efficacy and safety of the test drug
17. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
18. Has received a live vaccine within 30 days prior to the first dose of study drug. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (eg, FluMist®) are live attenuated vaccines and are not allowed.
19. Any history or presence of poorly controlled gastrointestinal disorders that could affect the absorption of the study drug (e.g. Crohn's disease, ulcerative colitis, chronic diarrhoea, malabsorption)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2019-01-24 (Actual); Primary Completion 2022-04-14 (Actual); Study Completion 2022-04-14 (Actual)

PRIMARY OUTCOMES:
Objective response rate | 2 years
  The objective response rate will be measured by RECIST 1.1.

SECONDARY OUTCOMES:
Overall survival | 2 years
  Overall survival: from the start of study treatment, to the time of death Progression free survival: from the start of study treatment, to the time of disease progression (RECIST 1.1) or death.
Toxicities | 2 years
  CTCAE 4.0, Grade 3 or higher

CONTACTS AND LOCATIONS:
Overall Officials: Ruey-Long Hong, MD PhD, Principal Investigator — Department of Oncology, National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Kao HF, Liao BC, Huang YL, Huang HC, Chen CN, Chen TC, Hong YJ, Chan CY, Chia JS, Hong RL. Afatinib and Pembrolizumab for Recurrent or Metastatic Head and Neck Squamous Cell Carcinoma (ALPHA Study): A Phase II Study with Biomarker Analysis. Clin Cancer Res. 2022 Apr 14;28(8):1560-1571. doi: 10.1158/1078-0432.CCR-21-3025. PMID 35046059